CLINICAL TRIAL: NCT06790004
Title: Endometrial Carcinoma: Comparison of Surgical Approaches (Laparoscopy vs Laparotomy) : Multicenter Retrospective Observational Study
Brief Title: Endometrial Carcinoma: Comparison of Surgical Approaches (Laparoscopy vs Laparotomy)
Acronym: LPSvsLPT
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 519/2020/OSS/AUSLRE
Record Dates: First submitted 2025-01-16; First posted 2025-01-23 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-01

CONDITIONS: Endometrial Carcinoma
Keywords: endometrial cancer; laparoscopy; laparotomy; minimally invasive surgery; risk of recurrence; Surgical complications
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Laparotomy; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with endometrial cancer who underwent surgical treatment: All patients with endometrial cancer who underwent surgical treatment from 2000 to 2020 at all participating centers in Emilia-Romagna.
  Interventions: Procedure: Laparotomy; Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparotomy — Open Surgery
Procedure: Laparoscopy — Minimally invasive surgery

SUMMARY:
Since the publication of the LAP2 study, a prospective randomized trial, laparoscopy has been considered the gold standard for treating patients with early-stage endometrial cancer (EC). However, no prospective randomized trials have been published reporting comparable data in patients with EC at high risk of recurrence (advanced stages or non-endometrioid histology). Nonetheless, some retrospective studies and a systematic review of the literature have demonstrated that minimally invasive surgery achieves better perioperative outcomes than laparotomy without compromising survival in patients with EC at high risk of recurrence.

The aim of this multicenter retrospective observational study is to evaluate the safety of minimally invasive surgery in treating EC at low, intermediate, and high risk of recurrence according to the ESMO-ESGO classification, based on cases treated in hospitals within the Emilia Romagna region. Specifically, we aim to assess the effects of a minimally invasive surgical approach compared to laparotomy in terms of:

1. Perioperative and postoperative complications: including the need for transfusions during and/or after surgery, duration of surgery, fever exceeding 38°C for more than 48 hours, and length of hospitalization.
2. Long-term oncological outcomes: including overall survival, disease-free survival, recurrence rates, recurrence sites, and time to recurrence.

This comparison will include patients treated for both endometrioid and non-endometrioid EC to provide a comprehensive evaluation of minimally invasive surgery versus laparotomy.

By delineating the safety and efficacy of laparoscopic techniques, particularly for higher-risk patients, this research could refine surgical standards and guide clinical decision-making, emphasizing evidence-based practices for tailored patient care. The study also aligns with broader efforts to optimize cancer management in regional and national healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of endometrial cancer who underwent surgical treatment between 2000 and 2020

Exclusion Criteria:

* Patients with other types of tumors (e.g., cervical or ovarian cancer).
* Patients for whom surgical and/or post-operative data are unavailable.
* Patients with a follow-up period of less than 6 months.
* Patients who refuse to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals assigned female at birth are eligible to participate in this study.
Study Population: Patients who underwent laparoscopic or laparotomic surgery for Type I or Type II endometrial cancer in the Emilia-Romagna region between 2000 and 2020
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Perioperative Complications | 30 days post-surgery.
  This metric assesses the number of participants with perioperative complications in the two intervention groups, specifically including the need for blood transfusions (either intraoperative or postoperative), surgery duration exceeding 180 minutes, postoperative fever >38°C lasting more than 48 hours, and hospitalization exceeding 7 days.

SECONDARY OUTCOMES:
Overall Survival (OS) | Five years post-surgery (from the date of surgery up to 5 years)
  Death from Any Cause
Disease-Free Survival (DFS) | Five years post-surgery (from the date of surgery up to 5 years)
  Time from Surgery to First Disease Recurrence or Death

OTHER OUTCOMES:
Pattern of recurrence | Five years post-surgery (from the date of surgery up to 5 years)
  Evaluation of the sites of recurrence, including pelvic relapse, lymph node relapse, and distant metastasis, with documentation of the timing of occurrence
Complete Cytoreduction | Time of surgery
  Assessment of complete surgical cytoreduction, defined as the absence of visible residual disease at the conclusion of surgery

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, RE
  - IRCCS - AOU Bologna, Bologna
  - Policlinico Sant'Orsola - Malpighi, Bologna
  - Azienda Ospedaliera- Universitaria Arcispedale Sant'Anna Ferrara, Ferrara
  - Ospedale Morgagni - Pierantoni, Forlì
  - Policlinico di Modena, Modena
  - AOU Parma, Parma
  - Ospedale di Rimini, AUSL Romagna, Rimini

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AIRTUM Working Group. I numeri del cancro in Italia 2015. http://www.registotumori.it/PDF/AIOM2015/I-numeri_del_cancro_2015.pd
- [Background] Papathemelis T, Oppermann H, Grafl S, Gerken M, Pauer A, Scharl S, Scharl A, Inwald E, Ignatov A, Ortmann O, Klinkhammer-Schalke M, Hein A, Beckmann MW, Lux MP. Long-term outcome of patients with intermediate- and high-risk endometrial cancer after pelvic and paraaortic lymph node dissection: a comparison of laparoscopic vs. open procedure. J Cancer Res Clin Oncol. 2020 Apr;146(4):961-969. doi: 10.1007/s00432-019-03122-8. Epub 2020 Jan 4. PMID 31901975
- [Background] Melamed A, Margul DJ, Chen L, Keating NL, Del Carmen MG, Yang J, Seagle BL, Alexander A, Barber EL, Rice LW, Wright JD, Kocherginsky M, Shahabi S, Rauh-Hain JA. Survival after Minimally Invasive Radical Hysterectomy for Early-Stage Cervical Cancer. N Engl J Med. 2018 Nov 15;379(20):1905-1914. doi: 10.1056/NEJMoa1804923. Epub 2018 Oct 31. PMID 30379613
- [Background] Ramirez PT, Frumovitz M, Pareja R, Lopez A, Vieira M, Ribeiro R, Buda A, Yan X, Shuzhong Y, Chetty N, Isla D, Tamura M, Zhu T, Robledo KP, Gebski V, Asher R, Behan V, Nicklin JL, Coleman RL, Obermair A. Minimally Invasive versus Abdominal Radical Hysterectomy for Cervical Cancer. N Engl J Med. 2018 Nov 15;379(20):1895-1904. doi: 10.1056/NEJMoa1806395. Epub 2018 Oct 31. PMID 30380365
- [Background] Scaletta G, Dinoi G, Capozzi V, Cianci S, Pelligra S, Ergasti R, Fagotti A, Scambia G, Fanfani F. Comparison of minimally invasive surgery with laparotomic approach in the treatment of high risk endometrial cancer: A systematic review. Eur J Surg Oncol. 2020 May;46(5):782-788. doi: 10.1016/j.ejso.2019.11.519. Epub 2019 Dec 2. PMID 31818527
- [Background] Papadia A, Garbade A, Gasparri ML, Wang J, Radan AP, Mueller MD. Minimally invasive surgery does not impair overall survival in stage IIIC endometrial cancer patients. Arch Gynecol Obstet. 2020 Feb;301(2):585-590. doi: 10.1007/s00404-019-05393-5. Epub 2019 Nov 28. PMID 31781888
- [Background] Walker JL, Piedmonte MR, Spirtos NM, Eisenkop SM, Schlaerth JB, Mannel RS, Spiegel G, Barakat R, Pearl ML, Sharma SK. Laparoscopy compared with laparotomy for comprehensive surgical staging of uterine cancer: Gynecologic Oncology Group Study LAP2. J Clin Oncol. 2009 Nov 10;27(32):5331-6. doi: 10.1200/JCO.2009.22.3248. Epub 2009 Oct 5. PMID 19805679
- [Background] Safdieh J, Lee YC, Wong A, Lee A, Weiner JP, Schwartz D, Schreiber D. A Comparison of Outcomes Between Open Hysterectomy and Robotic-Assisted Hysterectomy for Endometrial Cancer Using the National Cancer Database. Int J Gynecol Cancer. 2017 Sep;27(7):1508-1516. doi: 10.1097/IGC.0000000000001034. PMID 29470186
- [Background] Mourits MJ, Bijen CB, Arts HJ, ter Brugge HG, van der Sijde R, Paulsen L, Wijma J, Bongers MY, Post WJ, van der Zee AG, de Bock GH. Safety of laparoscopy versus laparotomy in early-stage endometrial cancer: a randomised trial. Lancet Oncol. 2010 Aug;11(8):763-71. doi: 10.1016/S1470-2045(10)70143-1. Epub 2010 Jul 16. PMID 20638901
- [Background] Ferguson SE, Panzarella T, Lau S, Gien LT, Samouelian V, Giede C, Steed H, Le T, Renkosinski B, Bernardini MQ. Prospective cohort study comparing quality of life and sexual health outcomes between women undergoing robotic, laparoscopic and open surgery for endometrial cancer. Gynecol Oncol. 2018 Jun;149(3):476-483. doi: 10.1016/j.ygyno.2018.04.558. Epub 2018 Apr 19. PMID 29681461
- [Background] Cancer Genome Atlas Research Network; Kandoth C, Schultz N, Cherniack AD, Akbani R, Liu Y, Shen H, Robertson AG, Pashtan I, Shen R, Benz CC, Yau C, Laird PW, Ding L, Zhang W, Mills GB, Kucherlapati R, Mardis ER, Levine DA. Integrated genomic characterization of endometrial carcinoma. Nature. 2013 May 2;497(7447):67-73. doi: 10.1038/nature12113. PMID 23636398
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231